CLINICAL TRIAL: NCT02735109
Title: Interest of the Confocal Microscope in the Diagnosis of Epidermoid Carcinoma of the Vulva and Their Precursors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: significant results after inclusion of 10 patients
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 14-AOI-13
Record Dates: First submitted 2015-03-17; First posted 2016-04-12 (Estimated); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Vulvar Mucosa Lesions; Vulvar Intraepithelial Neoplasia
Keywords: VIN
MeSH Terms: interventions — Photography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- description (Other): photographies and biopsy on normal area
  Interventions: Other: photographies; Procedure: biopsy normal area

INTERVENTIONS:
Other: photographies — cells description by taken photographies vith confocal microscope (VivaScope 3000)
Procedure: biopsy normal area — biopsy done to compare with abnormal area

SUMMARY:
The confocal microscope is a noninvasive imaging technique that provides high-resolution images to a depth of 250 microns, such as "optical" cuts in three dimensions in the thickness of the skin.

This is a single-center prospective descriptive study at the University Hospital of Nice in gynecology and dermatology.

The aim of the study is to describe the characteristics reproducibly for confocal microscope of normal vulvar mucosa lesions VIN, and vulvar squamous carcinoma.

The patients seen in consultation with vulvar lesions suspicious looking will be included.

The results will be compared systematically to the histological results of biopsies of lesions (gold standard).

DETAILED DESCRIPTION:
The squamous cell carcinoma is the most common cancer of the vulva (90-95%), with a prognosis depending on the stage. The management of vulvar intraepithelial neoplasia (VIN) is a secondary prevention of squamous cell carcinoma of the vulva.

Conventional VIN strongly associated with infection with oncogenic HPV (human papillomavirus) , present a risk of malignant degeneration of the order of 9-15%. Whereas the differentiated VIN, rarer often seen in the context of lichen sclerosis have a high risk of malignant degeneration ranging from 40 to 50%.

The diagnosis is histological, biopsy realization is currently the gold standard before starting a cure. However, biopsies on the vulva are not a harmless act for patients, and are often repeated due to extensive damage. The early management of lesions VIN avoids changes in squamous cell carcinoma. Over their diagnosed early, the better the care and specific treatments allocated.

The confocal microscope is a new imaging technology, already widely used for examination of the skin and mucous membranes. This is a noninvasive imaging technique that provides high-resolution images to a depth of 250 microns, such as "optical" cuts in three dimensions in the thickness of the skin. The device will be used for this study is the VivaScope 3000.

The advantage of the confocal microscope to discriminate between benign and malignant lesions of the skin and the oral mucosa has been shown in several prospective studies. Two recent studies have highlighted the promising results of the use of the confocal microscope for pigmented vulvar lesions (melanosis / melanoma).

There is currently no data in the literature on the impact of this technique on the VIN and vulvar epidermoid carcinomas.

This is a single-center prospective descriptive study at the University Hospital of Nice in gynecology and dermatology, to prove the contribution of the confocal microscope in vulvar intraepithelial neoplasia (VIN) and vulvar epidermoid carcinomas.

The aim of the study is to describe the characteristics reproducibly confocal microscope of normal vulvar mucosa lesions VIN, and vulvar squamous carcinoma.

The patients seen in consultation in the obstetrics and gynecology department and / or dermatology with a bow or vulvar lesions suspicious looking will be included in the study after signing an informed consent.

The results will be compared systematically to the histological results of biopsies of lesions (gold standard).

The investigators expect for this study a validation of the confocal microscope as a noninvasive diagnostic tool suspicious vulvar lesions (reduction of repeated biopsies, targeted biopsies to monitor certain lesions, and this even reduce health costs inherent to unnecessary biopsies)....

ELIGIBILITY:
Inclusion Criteria:

* Age = 18 years, Female
* Patient seen in consultation in the service of gynecology obstetrics, and, of dermatology of the Bow presenting during the medical examination one or several suspicious-looking vulvar hurts, suggestive of hurts of VIN or of carcinoma epidermoid vulvar
* Membership health secure
* Informed consent and paper of the obtained patient

Exclusion Criteria:

* Patient having already received a local treatment(processing) for hurts of VIN
* Pregnant Woman
* Patient under guardianship
* Not signature of the written consent and/or mental deficiency of the subject making its participation on approval impossible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Caracteristics of thorny layer, of granular layer,of basal layer of normal vulvar mucosa lesions VIN, and vulvar squamous cell carcinoma with confocal microscope | 12 months

SECONDARY OUTCOMES:
Caracteristics of thorny layer, of granular layer,of basal layer of normal vulvar mucosa lesions VIN, and vulvar squamous cell carcinoma with histological method | 12 months
Caracteristics of thorny layer, of granular layer,of basal layer of vulvar mucosa lesions VIN to descriptions and the observations of with the normal mucosa | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France